CLINICAL TRIAL: NCT01512329
Title: Pacing Activity Self-management for Patients With Multiple Sclerosis: Randomized Controlled Clinical Trial
Brief Title: Pacing Activity Self-management for Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University Hospital, Antwerp (Other); Universiteit Antwerpen (Other); Artesis University College, Antwerp (Other)
Responsible Party: Principal Investigator, Jo Nijs, associate professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PaceMS; Artesis University College (Other: Artesis University College Antwerp PWO)
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: neurology; physiotherapy; physical therapy; occupational therapy; stress management; activity management; treatment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pacing (Experimental): The pacing self-management program (3 one-on-one sessions weekly for 3 consecutive weeks) focused on teaching the patient to estimate their current physical capabilities prior to commencing an activity. In order to appropriately pace activities (daily activities and exercise bouts), MS patients were learned to estimate their current physical capabilities prior to commencing an activity, keeping in mind the regular fluctuating nature of their symptoms. The activity duration used within the program was less than that reported by the patient so to account for typical overestimations made by the patient. Each activity block was interspersed with breaks, with the length of this break equating to the duration of the activity.
  Interventions: Behavioral: pacing
- relaxation (Active Comparator): Relaxation therapy (3 one-on-one sessions weekly for 3 consecutive weeks) comprised of education about the role of stress in MS biology, and the opportunities stress management provides to handle this issue. Patients were then taught how to apply stress management techniques like Jacobson relaxation skills, Schultz relaxation skills, visualization, etc.
  Interventions: Behavioral: relaxation

INTERVENTIONS:
Behavioral: pacing — 3 one-on-one sessions weekly for 3 consecutive weeks
  Other Names: activity self-management; activity management
  Arms: pacing
Behavioral: relaxation — 3 one-on-one sessions weekly for 3 consecutive weeks
  Other Names: Schultz relaxation; visualisation; Jacobson relaxation; stress management
  Arms: relaxation

SUMMARY:
Given the lack of evidence in support of pacing self-management for patients with musltiple sclerosis (MS), it is examined whether physical behavior and health status of patients with MS improve in response to a pacing self-management program. The effects of pacing will be compared with those observed when applying relaxation therapy to patients with MS.

DETAILED DESCRIPTION:
Up to 50 patients fulfilling the criteria for the diagnosis of multiple sclerosis (MS) will be randomized to either 3 weeks of pacing activity self-management or relaxation therapy. Both treatment groups will receive 3 weekly sessions spread over 3 consecutive weeks. All treatments will be delivered by occupational therapists or physiotherapists. One treatment session lasts for about 45 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* adult
* age range between 18 and 65 years of age
* willing to sign informed consent form
* fulfilling the criteria for the diagnosis of multiple sclerosis

Exclusion Criteria:

- Not fulfilling each of the inclusion criteria listed above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the change in scores obtained from the Canadian Occupational Performance Measure (COPM) | measured at baseline (week 1) and post-treatment (week 5)
  Semi-structered interview.

SECONDARY OUTCOMES:
the change in subscale scores on the Medical Outcomes Short Form 37 Health Status Survey (SF-36) | measured once at baseline and once post-treatment
  The SF-36 assesses functional status and well-being or quality of life. The SF-36 has been documented to have reliability and validity in a wide variety of patient populations.
the change in subscale scores on the Checklist Individual Strength (CIS) | measured once at baseline and once post-treatment
  The CIS aims at assessing the subjective fatigue experience, concentration difficulties, motivation and physical activity. Higher scores on the CIS correspond to severe fatigue, many concentration difficulties, problems with motivation and a low level of physical activity. Its psychometric properties are well established.
the change in autonomic activity at rest and following 3 activities of daily living | measured once at baseline and once post-treatment
  The 3 activities of daily living entail writing a standardized test on a laptop computer, ironing, and climbing 26 flights of stairs. For measuring autonomic activity, the Nexus 10 device (Mind Media, the Netherlands) will be used. Skin conductance, body temperature, heart rate, blood volume pressure and heart rate variability will be measured continuously in real time during a 2 minutes period, with the patient sitting on a chair (back supported and hands resting on legs). Electrodes will be placed on the left hand in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Principal Investigator — Artesis University College, Antwerp; Daphne Kos, PhD, Study Director — Artesis University College, Antwerp
Locations (1):
- Nationaal Multiple Sclerosis Centrum, Melsbroek, Belgium

REFERENCES:
- [Background] Kos D, Nagels G, D'Hooghe MB, Duquet W, Ilsbroukx S, Delbeke S, Kerckhofs E. Measuring activity patterns using actigraphy in multiple sclerosis. Chronobiol Int. 2007;24(2):345-56. doi: 10.1080/07420520701282364. PMID 17453852
- [Background] Kos D, Nagels G, D'Hooghe MB, Duportail M, Kerckhofs E. A rapid screening tool for fatigue impact in multiple sclerosis. BMC Neurol. 2006 Aug 17;6:27. doi: 10.1186/1471-2377-6-27. PMID 16916440
- [Background] Kos D, Duportail M, D'hooghe M, Nagels G, Kerckhofs E. Multidisciplinary fatigue management programme in multiple sclerosis: a randomized clinical trial. Mult Scler. 2007 Sep;13(8):996-1003. doi: 10.1177/1352458507078392. Epub 2007 Jul 10. PMID 17623738
- See also: International Pain in Motion research group — http://www.paininmotion.be